CLINICAL TRIAL: NCT01136096
Title: Effects of Exercise Behavior Modification on Plasma Adiponectin and Insulin Resistance in High Risk Subjects of Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Ying-Tai Wu/, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 9261701067; DOH93-HP-1105 (Other Grant/Funding Number: Taiwan: Department of Health); DOH94-HP-1105 (Other Grant/Funding Number: Taiwan: Department of Health)
Record Dates: First submitted 2010-05-23; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; physical activity; adiponectin; metabolic risks; exercise; primary prevention
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): To promote participants' exercise behaviors with individualized home-based exercise program was designed based on the Health Belief Model and Transtheoretical Model
  Interventions: Behavioral: Physical activity promoting intervention
- Control (Other): Received oral instruction and written general education information without individualized exercise program
  Interventions: Behavioral: General instruction and education

INTERVENTIONS:
Behavioral: Physical activity promoting intervention — 1. An interview with a physiotherapist
  2. An exercise video specially designed by this study including warm-up, aerobic, cool-down and stretching exercises, and/or a simple exerciser to use at home
  3. An individualized home-based exercise program based on the Health Belief Model and Transtheoretical Model
  4. The daily record to check their body weight, exercise mode and duration
  5. Proper diet, caloric intake calculation, metabolic risk factors and prevention of diabetes were taught and a guide book was provided that included all the above mentioned details
  6. Telephone reminders of healthy lifestyle including the ways of overcoming barriers of regular exercise every 1 to 2 weeks for 3 months, 1-2 calls a month afterwards and no calls for the last month on a tapered off schedule
  Other Names: Home-based exercise; Exercise behavior modification
  Arms: Lifestyle counseling
Behavioral: General instruction and education — 1. Oral instruction and written general education information about weight control, proper diet and regular exercise in a one-page education brochure that was similar to the way used in the outpatient clinic
  2. Telephone reminders of healthy lifestyle every 1 to 2 weeks for 3 months, 1-2 calls a month afterwards and no calls for the last month on a tapered off schedule
  3. Without individualized exercise program and interview with a physiotherapist
  Other Names: General advice; Medical education
  Arms: Control

SUMMARY:
Investigators hypothesized home-based exercise intervention was beneficial to those who have had diabetic risk factor for type 2 diabetes mellitus

DETAILED DESCRIPTION:
This randomized clinical trial was designed to investigate whether a home-based exercise could improve adiponectin levels, exercise behavior and metabolic risk factors (insulin resistance, metabolic components and physical fitness) in subjects with at least a diabetic risk factor for type 2 diabetes mellitus. Participants were randomly allocated to either a control group or a home-based exercise group. All participants were evaluated for outcome measures at baseline, and at 3-month 6-month and 9-month follow-up after engaging in the intervention.

ELIGIBILITY:
Inclusion criteria:

* At least one of the following criteria as following: BMI >=24 kg/m*m, hypertension, dyslipidemia, fist-degree relatives of parents with type 2 diabetes, impaired glucose tolerance, gestational diabetes and delivering a babt weighing >=4.0 kg
* Ability of understanding Chinese or Taiwanese

Exclusion Criteria:

* Diabetes
* Receiving treatment with insulin or oral hypoglycemic agents
* Any other serious illness that prohibit them to undertake fitness evaluation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2004-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Plasma adiponectin level in μg/ml | Nine months after the start of the intervention
  Fasting blood samples were centrifuged to obtain plasma and then immediately stored at -20℃. Plasma adiponectin levels were then determined through enzyme-linked immunoassay (ELISA).
Exercise behavior | Nine months after the start of the intervention
  1. Exercise self-efficacy: Measured by exercise self-efficacy questionnaire in score
  2. Physical activity: Meausred by 7-day recall questionnaire in kcal/kg/day

SECONDARY OUTCOMES:
Insulin resistance | Three, 6 and 9 months after the start of the intervention
  plasma inulin level (μU/ml) meausred by AxSYM with HOMA-IR was caculated
Metabolic components | Three, 6 and 9 months after the start of the intervention
  1. Waist circumference (cm)
  2. Fasting blood samples were centrifuged to obtain plasma for plasma triglycerides (TG) and high-density lipoprotein (HDL) levels in mg/dl
  3. Plasma fasting glucose (FG) levels were measured in mg/dl by using the glucose oxidase membrane/hydrogen peroxide electrode method with the Antsense II analyzer (Bayer-Sankyo Co., Tokyo, Japan)
  4. Systolic blood pressure (SBP) and dystolic blood pressure (DBP) in mmHg
Physical fitness | Three, 6 and 9 months after the start of the intervention
  1. Body composition (kg/m^2): Body mass index that was weight in kilograms divided by the square of height in meter
  2. Flexibility (cm): Meausred by sit-and-reach test
  3. Grip strength (Nm): Measured by Jamar handheld dynameter
  4. Muscle endurance (times/min): Measured by sit-up test
  5. Cardiopulmonary fitness (3-minute step test)
Dietary intake | Three, 6 and 9 months after the start of the intervention
  Measured by 24-hour recall guestionnaire in kcal/kg/day
Plasma adiponectin level in μg/ml | Three and 6 months after the start of the intervention
  Fasting blood samples were centrifuged to obtain plasma and then immediately stored at -20℃. Plasma adiponectin levels were then determined through enzyme-linked immunoassay (ELISA)
Exercise behavior | Three and 6 months after the start of the intervention
  1. Exercise self-efficacy: Measured by exercise self-efficacy questionnaire in score
  2. Physical activity: Meausred by 7-day recall questionnaire in kcal/kg/day

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Doctor, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Esposito K, Pontillo A, Di Palo C, Giugliano G, Masella M, Marfella R, Giugliano D. Effect of weight loss and lifestyle changes on vascular inflammatory markers in obese women: a randomized trial. JAMA. 2003 Apr 9;289(14):1799-804. doi: 10.1001/jama.289.14.1799. PMID 12684358
- [Background] Arita Y, Kihara S, Ouchi N, Takahashi M, Maeda K, Miyagawa J, Hotta K, Shimomura I, Nakamura T, Miyaoka K, Kuriyama H, Nishida M, Yamashita S, Okubo K, Matsubara K, Muraguchi M, Ohmoto Y, Funahashi T, Matsuzawa Y. Paradoxical decrease of an adipose-specific protein, adiponectin, in obesity. Biochem Biophys Res Commun. 1999 Apr 2;257(1):79-83. doi: 10.1006/bbrc.1999.0255. PMID 10092513
- [Background] Hotta K, Funahashi T, Arita Y, Takahashi M, Matsuda M, Okamoto Y, Iwahashi H, Kuriyama H, Ouchi N, Maeda K, Nishida M, Kihara S, Sakai N, Nakajima T, Hasegawa K, Muraguchi M, Ohmoto Y, Nakamura T, Yamashita S, Hanafusa T, Matsuzawa Y. Plasma concentrations of a novel, adipose-specific protein, adiponectin, in type 2 diabetic patients. Arterioscler Thromb Vasc Biol. 2000 Jun;20(6):1595-9. doi: 10.1161/01.atv.20.6.1595. PMID 10845877
- [Background] Ouchi N, Kihara S, Arita Y, Maeda K, Kuriyama H, Okamoto Y, Hotta K, Nishida M, Takahashi M, Nakamura T, Yamashita S, Funahashi T, Matsuzawa Y. Novel modulator for endothelial adhesion molecules: adipocyte-derived plasma protein adiponectin. Circulation. 1999 Dec 21-28;100(25):2473-6. doi: 10.1161/01.cir.100.25.2473. PMID 10604883
- [Background] King H, Kriska AM. Prevention of type II diabetes by physical training. Epidemiological considerations and study methods. Diabetes Care. 1992 Nov;15(11):1794-9. doi: 10.2337/diacare.15.11.1794. PMID 1468317
- [Background] Li S, Shin HJ, Ding EL, van Dam RM. Adiponectin levels and risk of type 2 diabetes: a systematic review and meta-analysis. JAMA. 2009 Jul 8;302(2):179-88. doi: 10.1001/jama.2009.976. PMID 19584347
- [Derived] Chen CN, Chuang LM, Korivi M, Wu YT. Home-based exercise may not decrease the insulin resistance in individuals with metabolic syndrome. J Phys Act Health. 2015 Jan;12(1):74-9. doi: 10.1123/jpah.2013-0284. Epub 2014 Feb 5. PMID 24509907